CLINICAL TRIAL: NCT00004188
Title: A Randomized Study of Purged Versus Unpurged Peripheral Blood Stem Cell Transplant Following Dose Intensive Induction Therapy for High Risk Neuroblastoma
Brief Title: Combination Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3973; COG-A3973 (Other: Children's Oncology Group); CCG-A3973 (Other: Children's Cancer Group); POG-A3973 (Other: Pediatric Oncology Group); CCG-39703 (Other: Children's Cancer Group); FHCRC-1631.00; CDR0000067429 (Other: Clinical Trials.gov)
Record Dates: First submitted 2000-01-21; First posted 2003-01-27 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; etoposide phosphate; Isotretinoin; Melphalan; Topotecan; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (unpurged PBSC collection) (Experimental): Induction-3 wks (cyclophosphamide day 0&1, doxorubicin hydrochloride & vincristine sulfate day 0-2 & filgrastim(G-CSF) day 3 crs 1,2,4 & 6.) Crs 3 & 5 (etoposide day 0-2, cisplatin day 0-3, G-CSF day 4). Pts undergo unpurged PBSC collection until the target cell count is reached. Surgical resection of the tumor after crs 5 of induct. CR, VGPR, PR after induct receive consolidation (melphalan day -7 to -5, carboplatin & etoposide day -7 to -4. purged peripheral blood stem cell transplantation infusion day 0, G-CSF 4 hrs post transplant. Day 66, isotretinoin 2x day/14 days. Isotretinoin every 4 wks 6 crs. After consol (28 days from stem cell infusion), radiation therapy 1x day/7 days. Not undergoing autologous bone marrow transplantation receive maintenance(cyclophosphamide 30 mins, topotecan hydrochloride days 0-4, G-CSF day 5). Maint every 3 wks/3 crs. Radiation therapy and Isotretinoin 2x day/14 days then every 4 wks for 6 crs.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cisplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: isotretinoin; Drug: melphalan; Drug: topotecan hydrochloride; Drug: vincristine sulfate; Procedure: autologous bone marrow transplantation; Procedure: bone marrow ablation with stem cell support; Procedure: conventional surgery; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy
- Arm II (unpurged PBSC collection) (Experimental): Induction-3 wks (cyclophosphamide day 0&1, doxorubicin hydrochloride & vincristine sulfate day 0-2 & filgrastim(G-CSF) day 3 crs 1,2,4 & 6.) Crs 3 & 5 (etoposide day 0-2, cisplatin day 0-3, G-CSF day 4). Immunocytology + PBSC undergo purged autologous bone marrow collection or repeat purged or unpurged PBSC collection. Surgical resection of the tumor after crs 5 of induct. CR, VGPR, PR after induct receive consolidation (melphalan day -7 to -5, carboplatin & etoposide day -7 to -4. Unpurged peripheral blood stem cell transplantation infusion day 0, G-CSF 4 hrs post transplant. Day 66, isotretinoin 2x day/14 days. Isotretinoin every 4 wks 6 crs. After consol (28 days from stem cell infusion), radiation therapy 1x day/7 days. Not undergoing autologous bone marrow transplantation receive maintenance(cyclophosphamide 30 mins, topotecan hydrochloride days 0-4, G-CSF day 5). Maint every 3 wks/3 crs. Radiation therapy and Isotretinoin 2x day/14 days then every 4 wks for 6 crs.
  Interventions: Drug: carboplatin; Drug: cisplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: isotretinoin; Drug: melphalan; Drug: topotecan hydrochloride; Drug: vincristine sulfate; Procedure: autologous bone marrow transplantation; Procedure: bone marrow ablation with stem cell support; Procedure: conventional surgery; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — Given IV
  Other Names: GRANULOCYTE COLONY-STIMULATING FACTOR; r-metHuG-CSF; G-CSF; Neupogen; NSC 614629
  Arms: Arm I (unpurged PBSC collection)
Drug: carboplatin — Given IV
  Other Names: Paraplatin; NSC #241240
Drug: cisplatin — Given IV
  Other Names: Cis-diamminedichloroplatinum II; Platinol-AQ; NSC #11987
Drug: cyclophosphamide — Given IV
  Other Names: CTX; Cytoxan; NSC #026271
Drug: doxorubicin hydrochloride — Given IV
  Other Names: Adriamycin; NSC #123127; IND #7038
Drug: etoposide — Given IV
  Other Names: VP-16; VePesid; Etopophos; NSC #141540
Drug: isotretinoin — Given IV
  Other Names: 13-cis-retinoic acid; RO-43; 780; Accutane; Amnesteem; Claravis; NSC 329481
Drug: melphalan — Given IV
  Other Names: L-phenylalanine mustard; phenylalanine mustard; L-PAM; L-sarcolysin; NSC 008806
Drug: topotecan hydrochloride — Given IV
  Other Names: SKF-104864; Hycamtin; NSC #609699
Drug: vincristine sulfate — Given IV
  Other Names: VCR; Oncovin; NSC #067574
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: conventional surgery — All patients undergo delayed surgical resection of the residual tumor after course 5 of induction chemotherapy
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy — After completion of consolidation (at least 28 days from stem cell infusion), all patients receive local radiotherapy daily over 7 days

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: This randomized phase III trial is studying peripheral stem cell transplantation with treated peripheral stem cells following combination chemotherapy to see how well it works compared to peripheral stem cell transplantation with untreated peripheral stem cells following combination chemotherapy in treating patients with neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the event-free survival in patients with newly diagnosed high risk neuroblastoma or ganglioneuroblastoma treated with myeloablative consolidation chemotherapy and autologous purged versus unpurged peripheral blood stem cells (PBSC).
* Compare the time to engraftment and CD34 content and tumor content by reverse transcriptase polymerase chain reaction (RT-PCR) of purged versus unpurged PBSC in patients treated with these regimens.
* Determine event-free survival of patients treated with dose intensive induction chemotherapy comprising cyclophosphamide, doxorubicin, and vincristine alternating with cisplatin and etoposide.
* Determine the toxicity of this dose-intensive induction chemotherapy regimen in these patients.
* Evaluate tumor resectability at second look or delayed surgery, response (complete response and very good partial response) at completion of induction therapy, tumor content of peripheral blood and bone marrow, and the comparison of historical data from CCG-3891 induction therapy in these patients.

Secondary

* Compare the toxicity of this myeloablative consolidation regimen using purged vs unpurged PBSC in these patients.
* Determine if event-free survival is predictable by RT-PCR positivity of the stem cell, minimal residual disease in bone marrow and peripheral blood after transplantation by immunocytology, and extent of disease as measured by MIBG after transplantation in patients treated with these regimens.
* Evaluate the prognostic impact of tumor biology on event free survival in patients treated with these regimens.
* Determine the incidence of relapse in the primary site after radiotherapy and in irradiated versus unirradiated metastatic sites in these patients.
* Assess the toxicity and tolerability of maintenance therapy with topotecan and cyclophosphamide after intensive induction therapy in patients who decline or are unable to receive myeloablative therapy.
* Determine the health-related quality of life of patients treated with these regimens.
* Compare late effects of these regimens on the growth, endocrine, pulmonary, and cardiac function of these patients vs general population standards.
* Determine the incidence of second malignant neoplasms in patients treated with these regimens.
* Determine the variability of isotretinoin pharmacokinetics and relationship to pharmacogenomic parameters in these patients.
* Correlate the isotretinoin pharmacokinetics and pharmacogenomic parameters and/or genetic variations in isotretinoin metabolic enzymes with event-free survival or systemic toxicity in these patients.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms for peripheral blood stem cell (PBSC) collection.

All patients receive induction chemotherapy comprising cyclophosphamide IV over 6 hours on days 0 and 1, doxorubicin IV and vincristine IV continuously over 72 hours on days 0-2, and filgrastim (G-CSF) subcutaneously (SC) or IV beginning on day 3 and continuing until blood counts recover for courses 1, 2, 4, and 6. Treatment alternates with courses 3 and 5 comprising etoposide IV over 2 hours on days 0-2, cisplatin IV over 1 hour on days 0-3, and G-CSF SC or IV beginning on day 4 and continuing until blood counts recover. Induction chemotherapy repeats every 3 weeks or when blood counts recover in the absence of disease progression or unacceptable toxicity.

After course 2 or 3 of induction chemotherapy, patients undergo PBSC collection, either purged or unpurged, depending on randomization. Patients continue on daily G-CSF until cell collection is complete.

* Arm I: Patients undergo unpurged PBSC collection until the target cell count is reached.
* Arm II: Patients undergo purged PBSC collection until the target cell count is reached.

Patients with immunocytology positive PBSC undergo purged autologous bone marrow collection or repeat purged or unpurged PBSC collection depending on individual patient characteristics.

All patients undergo delayed surgical resection of the residual tumor after course 5 of induction chemotherapy.

After induction therapy, patients achieving complete response, very good partial response, or partial response receive consolidation therapy comprising melphalan IV on days -7 to -5 followed by carboplatin IV and etoposide IV continuously over days -7 to -4. Patients receive purged or unpurged PBSC infusion or purged autologous bone marrow transplantation on day 0 followed by G-CSF SC or IV beginning 4 hours after completion of transplantation and continuing until blood counts recover. Beginning on day 66, patients receive oral isotretinoin twice daily for 14 days. Isotretinoin therapy repeats every 4 weeks for 6 courses.

After completion of consolidation (at least 28 days from stem cell infusion), all patients receive local radiotherapy daily over 7 days.

Patients not undergoing transplantation or who are ineligible for consolidation therapy receive maintenance therapy comprising cyclophosphamide IV over 30 minutes followed by topotecan IV over 30 minutes on days 0-4. Patients receive G-CSF SC or IV beginning on day 5 and continuing until blood counts recover. Maintenance therapy repeats every 3 weeks for 3 courses. After completion of maintenance therapy, patients receive radiotherapy as outlined above. Patients then receive oral isotretinoin twice daily for 14 days. Isotretinoin therapy repeats every 4 weeks for 6 courses.

Quality of life is assessed at 1* and 5 years.

Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually thereafter or until disease progression.

NOTE: * Patients under 5 years of age at 1 year are not assessed until 5 years.

PROJECTED ACCRUAL: A total of 486 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed neuroblastoma OR ganglioneuroblastoma, and/or evidence of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites, meeting 1 of the following criteria:

  * Age greater than 18 months with stage IV disease, regardless of biologic factors
  * Age 12-18 months with stage IV disease meeting one of the following criteria:

    * Any unfavorable biologic feature (e.g., MYCN amplification, unfavorable pathology, and/or DNA index = 1)
    * Any biologic feature that is indeterminate, unsatisfactory, or unknown
* At least 1 year old with the following:

  * Stage IIa/IIb with MYCN amplification (> 10) AND unfavorable pathology
  * Stage III with MYCN amplification (> 10) OR unfavorable pathology
  * Stage I, II, or IVS with disease progression to stage IV without interval chemotherapy

    * No more than 3 weeks since progression
    * Must have been enrolled on protocol CCG-B973, COG-ANBL00B1, or POG-9047
* Less than 1 year old with the following:

  * Stage III, IV, or IVS disease with MYCN amplification (> 10)
* Registration on protocol COG-ANBL00B1 required within 14 days of diagnosis

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics
* 30 and under at time of diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Inadequate hematopoiesis secondary to bone marrow involvement with > 10% tumor infiltration allowed

Hepatic:

* Bilirubin ≤ 1.5 mg/dL
* ALT ≤ 300 units/L

Renal:

* Creatinine ≤ 1.5 mg/dL
* Creatinine clearance or glomerular filtration rate ≥ 60 mL/min

Cardiovascular:

* ECG normal
* Ejection fraction ≥ 55% by echocardiogram or MUGA OR
* Fractional shortening ≥ 28% by echocardiogram

Other:

* Able to tolerate peripheral blood stem cell collection
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for at least 1 month prior to, during, and for 1 month after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No more than 1 prior course of chemotherapy on the Intergroup low/intermediate risk neuroblastoma study (P9641, A3961)

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior localized emergency radiotherapy to sites of life-threatening or function-threatening disease allowed

Surgery:

* Not specified

Other

* No other prior systemic therapy

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 495 (Actual)
Dates: Start 2001-02; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Event-free survival rate | Time from study registration until the time of the first occurrence of either relapse, progression, secondary malignancy, or death, or until the time of last contact with the patient if none of these events occurs, assessed up to 6 years
Rate of occurrence of toxic (non disease-related) deaths where a toxic death will be "counted" if it occurs prior to the initiation of the immunotherapy | Up to day 42

SECONDARY OUTCOMES:
Time to engraftment | Up to 6 years
  Engraftment is defined as three consecutive measurements of ANC > 500.
CD34 content | Up to 6 years
Tumor content as measured by reverse transcriptase polymerase chain reaction | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan G. Kreissman, MD, Study Chair — Duke Cancer Institute
Locations (96):
- United States (86):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - University of Illinois at Chicago Cancer Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan, Ann Arbor, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospital of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Background] Dubois SG, Geier E, Batra V, Yee SW, Neuhaus J, Segal M, Martinez D, Pawel B, Yanik G, Naranjo A, London WB, Kreissman S, Baker D, Attiyeh E, Hogarty MD, Maris JM, Giacomini K, Matthay KK. Evaluation of Norepinephrine Transporter Expression and Metaiodobenzylguanidine Avidity in Neuroblastoma: A Report from the Children's Oncology Group. Int J Mol Imaging. 2012;2012:250834. doi: 10.1155/2012/250834. Epub 2012 Sep 25. PMID 23050139
- [Background] Cantos MF, Gerstle JT, Irwin MS, Pappo A, Farley S, Cheang T, Kim PC. Surgical challenges associated with intensive treatment protocols for high-risk neuroblastoma. J Pediatr Surg. 2006 May;41(5):960-5. doi: 10.1016/j.jpedsurg.2006.01.059. PMID 16677893
- [Background] Kushner BH, Budnick A, Kramer K, Modak S, Cheung NK. Ototoxicity from high-dose use of platinum compounds in patients with neuroblastoma. Cancer. 2006 Jul 15;107(2):417-22. doi: 10.1002/cncr.22004. PMID 16779793
- [Result] Landier W, Knight K, Wong FL, Lee J, Thomas O, Kim H, Kreissman SG, Schmidt ML, Chen L, London WB, Gurney JG, Bhatia S. Ototoxicity in children with high-risk neuroblastoma: prevalence, risk factors, and concordance of grading scales--a report from the Children's Oncology Group. J Clin Oncol. 2014 Feb 20;32(6):527-34. doi: 10.1200/JCO.2013.51.2038. Epub 2014 Jan 13. PMID 24419114
- [Result] Naranjo A, Parisi MT, Shulkin BL, London WB, Matthay KK, Kreissman SG, Yanik GA. Comparison of (1)(2)(3)I-metaiodobenzylguanidine (MIBG) and (1)(3)(1)I-MIBG semi-quantitative scores in predicting survival in patients with stage 4 neuroblastoma: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2011 Jul 1;56(7):1041-5. doi: 10.1002/pbc.22991. Epub 2011 Feb 15. PMID 21328522
- [Result] Yanik GA, Parisi MT, Naranjo A, et al.: MIBG scoring as a prognostic indicator in patients with stage IV neuroblastoma: A COG study. [Abstract] J Clin Oncol 28 (Suppl 15): A-9516, 2010.
- [Result] Kreissman SG, Villablanca JG, Diller L, et al.: Response and toxicity to a dose-intensive multi-agent chemotherapy induction regimen for high risk neuroblastoma (HR-NB): a Children's Oncology Group (COG A3973) study. [Abstract] J Clin Oncol 25 (Suppl 18): A-9505, 527s, 2007.
- [Derived] Kreissman SG, Seeger RC, Matthay KK, London WB, Sposto R, Grupp SA, Haas-Kogan DA, Laquaglia MP, Yu AL, Diller L, Buxton A, Park JR, Cohn SL, Maris JM, Reynolds CP, Villablanca JG. Purged versus non-purged peripheral blood stem-cell transplantation for high-risk neuroblastoma (COG A3973): a randomised phase 3 trial. Lancet Oncol. 2013 Sep;14(10):999-1008. doi: 10.1016/S1470-2045(13)70309-7. Epub 2013 Jul 25. PMID 23890779